CLINICAL TRIAL: NCT00407433
Title: Phase 2 Single-Arm Studies of Gemcitabine in Combination With Oxaliplatin Refractory and Relapsed Pediatric Solid Tumors
Brief Title: Clinical Studies of Gemcitabine-Oxaliplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGR 1205; ITCC-004-GEMOX
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Medulloblastoma; Central Nervous System Tumors; Neuroblastoma; Osteosarcoma
Keywords: Gemcitabine; Oxaliplatine; Paediatric solid tumors; Other CNS tumors; Other miscellaneous solid non-CNS tumours
MeSH Terms: conditions — Medulloblastoma; Central Nervous System Neoplasms; Neuroblastoma; Osteosarcoma | interventions — Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine (Gemzar®), Oxaliplatin (Eloxatin®)

SUMMARY:
These are Phase 2 single-arm studies of gemcitabine in combination with oxaliplatin in refractory or relapsing pediatric solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant solid tumor (at diagnosis)
* Relapsed or refractory tumors in which correct standard treatment approaches have failed
* Measurable primary and/or metastatic disease: at least one bi-dimensionally measurable lesion. For patients with neuroblastoma, measurable disease will be defined by the modified International Neuroblastoma Staging System (Brodeur et al.1993). For patients with osteosarcoma, measurable lesions are lung metastases and osseous lesions with soft tissue tumor, in exclusion of completely calcified or necrosed lesion at study entry. A patient with an unique osseous lesion without soft tissue mass can be included in the study if the lesion is operable and thus accessible for histological response assessment.
* No more than one salvage therapy for relapse
* Age at inclusion: 6 months to ≤ 20 years
* Lansky play score ≥ 70% or ECOG performance status ≤ 1
* Life expectancy ≥ 3 months
* Adequate organ function:

  * Adequate hematological function: neutrophil count >= 1.0 x 10^9/L, platelet count >= 100 x 10^9/L; in case of bone marrow disease: >= 75 x 10^9/L; hemoglobin >= 8 g/dL
  * Adequate renal function: creatinine > 1.5 x ULN for age; If serum creatinine is > 1.5 ULN of age, then creatinine clearance (or radioisotope GFR) must be > 70 ml/min/1.73 m2 Adequate hepatic function: bilirubin > 1.5 x ULN; AST and ALT > 2.5 x ULN (AST, ALT ≤ 5 x ULN in case of liver metastases).
* Wash out of 3 weeks in case of prior chemotherapy, 6 weeks if treatment included nitrosoureas, 2 weeks in case of vincristine alone; 4 weeks in case of prior radiotherapy. Patients must have recovered from the acute toxic effects of all prior therapy before enrollment into the study.
* Able to comply with scheduled follow-up and with management of toxicity
* All patients with reproductive potential must practice an effective method of birth control while on study. Female patients with childbearing potential must have a negative pregnancy test within 7 days before study treatment.
* Written informed consent from patient, parents or legal guardian

Exclusion Criteria:

* Concurrent administration of any other antitumor therapy.
* Have previously completed or withdrawn from this study or any other study investigating gemcitabine or oxaliplatin.
* Have a serious concomitant systemic disorder (for example, active infection including HIV or cardiac disease) that in the opinion of the investigator, would compromise the patient's ability to complete the study
* Pre-existing sensory or motor neuropathy >Grade 2 (excluding neuropathy due to disease and/or surgery)
* History of allergic reaction to platinum compounds
* Are pregnant or breast feeding
* Presence of symptomatic brain metastases in patients with solid non-central nervous system (CNS) tumors

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint for efficacy is the percentage of patients achieving complete or partial response according to WHO guidelines, after having received 4 cycles of gemcitabine-oxaliplatin (8 weeks).

SECONDARY OUTCOMES:
The secondary efficacy variables are the duration of response, the time to treatment failure, the time to progressive disease and the overall survival.
Clinical and laboratory toxicities/symptomatology will be graded according to NCI-Common toxicity criteria AE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Geoerger, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France